CLINICAL TRIAL: NCT04223908
Title: InFocus France Epidemiological Study of Health Burden in Major Hypertriglyceridemia
Acronym: InFocus
Status: Completed | Type: Observational
Sponsor: New French Society of Atherosclerosis (Other)
Collaborators: Akcea Therapeutics (Industry)
Responsible Party: Principal Investigator, Philippe Moulin, Clinical professor / head department of endocrinology, Hospices Civils de Lyon
Other Study IDs: 2018-A01735-50
Record Dates: First submitted 2020-01-02; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Familial Chylomicronemia Syndrome; Multifactorial Chylomicronemia Syndrome
Keywords: major hypertriglyceridemia; health burden
MeSH Terms: conditions — Familial hyperchylomicronemia syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FCS: patient with genetically documented familial chylomicronemia syndrome
  Interventions: Other: observational : questionnaries for assessment of health burden
- MCS: patient with genetically or phenotypically documented multifactorial chylomicronemia syndrome
  Interventions: Other: observational : questionnaries for assessment of health burden

INTERVENTIONS:
Other: observational : questionnaries for assessment of health burden — The French IN-FOCUS study was designed to capture current and retrospective data in FCS or MCS. Patients were called by the participating centers and were proposed to answer a paper questionnaire or to connect to a web-based questionnaire The questionnaire was divided into sections specifically assessing various domains of their experience: demographic data, signs, symptoms and complications of the disease, healthcare circuit, management, relationship with healthcare providers, and burden of the disease on daily life. (Details are available as supplementary material S1). The questionnaire focused on symptoms because the interest of quality of life assessment tools is debated in rare diseases with episodic manifestations. Indeed, most of these tools refer to a limited recall period.

SUMMARY:
FCS and MCS patients recruited from 7 academic reference centers were invited to answer a paper or a web questionnaire. Questions encompassed demographics, physical, cognitive and mental symptoms, health care circuit, past and current disease management, satisfaction regarding healthcare providers and impact on daily life.

DETAILED DESCRIPTION:
cross-sectional study involving a sample of FCS and MCS patients in 1:1 ratio. The study was run in seven academic reference centers in France. Adult patients with documented history of fasting TG > 10 mmol/L (885 mg/dL) were recruited. Patients had to be genetically characterized or MCS patients had a MCS score ≤ 9 [11]. Group sample sizes of 19 FCS and 19 MCS have been calculated to achieve an at least 80% power to detect a 40% difference in the frequency of abdominal pain assuming that 90% of FCS patients would complain about abdominal pain.

The study protocol was approved by a nationally appointed ethics committee (Comité de Protection des Personnes - Ile de France 5) under number 18040. The study protocol complied with the ethical guidelines of the Declaration of Helsinki and the French Bioethics Law Jarde. The data management complied with the CNIL requirement. Each patient was informed about the aims and constraints of the study and signed a non-opposition form prior to any study procedure.

Health Burden assessment The French IN-FOCUS study was designed to capture current and retrospective data in FCS or MCS. Patients were called by the participating centers and were proposed to answer a paper questionnaire or to connect to a web-based questionnaire The questionnaire was divided into sections specifically assessing various domains of their experience: demographic data, signs, symptoms and complications of the disease, healthcare circuit, management, relationship with healthcare providers, and burden of the disease on daily life. (Details are available as supplementary material S1). The questionnaire focused on symptoms because the interest of quality of life assessment tools is debated in rare diseases with episodic manifestations. Indeed, most of these tools refer to a limited recall period.

Data analysis The statistical analysis was performed by Soladis (Lyon, France) using the Statistical Analysis System (SAS) software 9.4 (SAS Institute, Cary, NC, USA). Continuous variables were summarized by the number of observed data, mean, standard deviation (SD), median, first and third quartiles. Categorical variables were described as numbers and percentages calculated on the number of observed data. FCS and MCS subjects were compared using Student's t test or U Mann-Whitney's test. Categorical variables were compared by the chi squared test or the Fisher's exact test. Tests were two-sided and the significance threshold was set at 5%. No adjustment of the Type 1 error risk was made for multiplicity. Impact of history of AP was evaluated in a multivariable model (logistic regression for binary variables, ordinal logistic regression for ordinal variables) including the type of disease (FCS or MCS), history of AP and the interaction between these two predictors.

ELIGIBILITY:
Inclusion Criteria:

* any adult FCS patient genetically documented any adult MCS patient genetically or phenotypically documented

Exclusion Criteria:

* legal restrictions

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: cross-sectional study involving a sample of FCS and MCS patients in 1:1 ratio. The study was run in seven academic reference centers in France. Adult patients with documented history of fasting TG > 10 mmol/L (885 mg/dL) were recruited. Patients had to be genetically characterized or MCS patients had a MCS score ≤ 9 [11]. Group sample sizes of 19 FCS and 19 MCS have been calculated to achieve an at least 80% power to detect a 40% difference in the frequency of abdominal pain assuming that 90% of FCS patients would complain about abdominal pain
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
abdominal pain | 12 previous months record
  Symptoms were assessed as present/absent within the 12 months prior to the study; if present, the patient was asked to rate their frequency (yearly, every 3 months, monthly, weekly, daily using a 5-point verbal numeric scale) and severity using a 7-point verbal numeric scale with 1=very mild and 7=very important.

SECONDARY OUTCOMES:
dietary burden | 12 previous months records
  Consuming more fats than allowed to avoid attracting attention Longing for rich-fat food Meals lack variety Carefully reading the food labelling Feeling frustrated by his/her diet Controlling fat consumption is a hard task Avoids alcohol consumption to prevent symptoms Fasting voluntarily Preparing a special meal different from the rest of the family
  Symptoms were assessed as present/absent within the 12 months prior to the study; if present, the patient was asked to rate their frequency (yearly, every 3 months, monthly, weekly, daily using a 5-point verbal numeric scale) and severity using a 7-point verbal numeric scale with 1=very mild and 7=very important.
psychological burden | 12 previous months record
  Feeling anxious when eating out Feeling anxious if not compliant with his/her diet Trouble concentrating due to insufficient satiety Feeling guilty when drinking small amounts of alcohol Symptoms were assessed as present/absent within the 12 months prior to the study; if present, the patient was asked to rate their frequency (yearly, every 3 months, monthly, weekly, daily using a 5-point verbal numeric scale) and severity using a 7-point verbal numeric scale with 1=very mild and 7=very important.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Moulin, Study Chair — New French Atherosclerosis Siciety
Locations (1):
- new French society of atherosclerosis, Saint-Maur-des-Fossés, France

IPD SHARING:
Plan to Share IPD: Yes
according agreement of PI, NSFA Board and complience with CNIL
Supporting Information: Study Protocol, SAP, ICF